CLINICAL TRIAL: NCT06194019
Title: Evaluation of Volume Status Changes in Children on Regular Hemodialysis at Assiut University Children,s Hospital
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Collaborators: Professor Mohamed mahrous Eltallawy (Unknown); Assistant Professor Ahlam Badawy Ali (Unknown); Lecturer Asmaa Ahmed Mahmoud (Unknown)
Responsible Party: Principal Investigator, Ahlam Abelbaset Mohamed, assistant lecturer, Assiut University
Other Study IDs: volume status
Record Dates: First submitted 2023-12-21; First posted 2024-01-08 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2023-12

CONDITIONS: Volume Status in Chronic Kidney Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: lung ultrasonography — N-terminal pro-brain natriuretic peptide (NT-proBNP) as a biomarker for detection volume overload.
  Other Names: Bioimpedance analysis (BIA)

SUMMARY:
Chronic kidney disease (CKD) is a major health problem worldwide.(1) Chronic renal failure is defined as a decrease in glomerular filtration rate (GFR) of less than 60 ml/min/1.73 m2 of body surface evolving for more than 3 months

DETAILED DESCRIPTION:
Chronic kidney disease (CKD) is a major health problem worldwide.(1) Chronic renal failure is defined as a decrease in glomerular filtration rate (GFR) of less than 60 ml/min/1.73 m2 of body surface evolving for more than 3 months . The etiologies of CKD in children are three main groups of pathologies: congenital anomalies of the kidney and urinary tract , hereditary nephropathies and acquired causes . (2) complication of pediatric hemodialysis is chronic fluid overload, left ventricular hypertrophy ,hypertension, heart failure, decrease arterial flexibility and often results in increase chance of morbidity and mortality, So fluid overload must be prevented .(3) Lung ultrasonography is the most recent, safe, easy, and reliable technique . The most commonly observed finding is a comet tail fanning out from the lung-wall interface and spreading upwards to the edge of the screen, named a "B-line" Chest sonar advantages include its noninvasiveness , ease of use, availability of portable machines, avoidance of radiation detect lung edema even in initial non symptomatic cases known as hidden lung congestion .(4) Bioimpedance analysis (BIA) Bio impedance spectroscopy (BIS) is a technique used to estimate total body water, extracellular water, lean and adipose tissue mass and over hydration . (5) N-terminal pro-brain natriuretic peptide is used as a biomarker to aid to predict cardiac dysfunction in children and adolescents .(6)it is an effective marker of volume status in patient with or without reduced ejection fraction undergoing hemodialysis. (7)

ELIGIBILITY:
Inclusion Criteria:

- Patients aged 3 to 16 years having end stage renal disease undergoing regular haemodialysis for at least more than 6 months of both gender were enrolled

Exclusion Criteria:

* Patients with chronic lung disease ,or pulmonary infection in the last 2 months were excluded from study.

Patients with congestive heart failure Patients with Pulmonary edema Patient with pericardial effusion parental refusal to participate

Ages: 3 Years to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: All cases with end stage renal diseases undergoing regular haemodialysis in nephrology department in a period of two year
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of volume status changes in children on regular hemodialysis at Assiut university children's hospital | two year
  Evaluation of Volume status in children on regular haemodialysis by Chest sonar Evaluation of Volume status in children on regular haemodialysis by Chest sonar
  Evaluation of Volume status in children on regular haemodialysis by Chest sonar
  Evaluation of Volume status in children on regular haemodialysis by Chest sonar Evaluation of Volume status in children on regular haemodialysis by Chest sonar

CONTACTS AND LOCATIONS:
Overall Officials: Ahlam Badawy, assist prof, Study Director — Assiut University; Asmaa Ahmed, lecturer, Study Director — Assiut University

IPD SHARING:
Plan to Share IPD: No